CLINICAL TRIAL: NCT01829048
Title: A Randomized, Double-blind, Placebo Controlled, Sponsor Open, Phase 1b Study To Examine The Adjunctive Safety, Tolerability And Pharmacokinetics Of Pf-02545920 In Psychiatrically Stable Subjects With Schizophrenia
Brief Title: A Study To Examine The Safety, Tolerability And Pharmacokinetics Of PF-02545920 In Psychiatrically Stable Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Basic Science
Other Study IDs: A8241018
Record Dates: First submitted 2013-03-06; First posted 2013-04-11 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2017-11

CONDITIONS: Schizophrenia
Keywords: PF-02545920; safety; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — 2-((4-(1-methyl-4-pyridin-4-yl-1H-pyrazol-3-yl)phenoxy)methyl)quinoline; KPNA1 protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PF-02545920 (Experimental)
  Interventions: Drug: PF-02545920
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-02545920 — 15 mg (2 mg X 2d, 5 mg X 2d, 8 mg X 3 d, then 15 mg) Q12h
  Other Names: Cohort 1
  Arms: PF-02545920
Drug: PF-02545920 — 15 mg (5 mg X 2d, 10 mg X 2d, then 15 mg) Q12h
  Other Names: Cohort 2
  Arms: PF-02545920
Drug: PF-02545920 — 15 mg (5 mg BID for 7 days 10 mg BID for 7 days, then 15 mg BID for 4 days) Q12h
  Other Names: Cohort 3
  Arms: PF-02545920
Drug: Placebo — Placebo Q12h
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of multiple doses of PF 02545920 administered orally to psychiatrically stable subjects with schizophrenia receiving background antipsychotic +/- other adjunctive medication.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatrically stable subjects with schizophrenia.
* Evidence of stable schizophrenia symptomatology greater than or equal to 3 months.
* Subjects must be on a stable medication treatment regimen greater than or equal to 2 months, including concomitant psychotropic medications.

Exclusion Criteria:

* History of seizures or of a condition with risk of seizures.
* Subjects who have had electroconvulsive therapy within the 6 months prior to randomization.
* Pregnant or nursing females, and females of child bearing potential.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2013-03-06 (Actual); Primary Completion 2013-10-17 (Actual); Study Completion 2013-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- California Clinical Trials Medical Group, Glendale, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-02545920 (Cohort 1): Participants received PF-02545920 15 milligram (mg) orally in a titrated manner over 10 days (titration scheme: 2 mg every 12 hours for 2 days, then 5 mg every 12 hours for 2 days, then 8 mg every 12 hours for 3 days, and then 15 mg every 12 hours for 3 days).
- PF-02545920 (Cohort 2): Participants received PF-02545920 15 mg orally in a titrated manner over 10 days (titration scheme: 5 mg every 12 hours for 2 days, then 10 mg every 12 hours for 2 days, and then 15 mg every 12 hours for 6 days).
- Placebo (Cohorts 1 and 2): Participants received placebo-matched to PF-02545920 tablets (Cohort 1 or 2) every 12 hours orally for 10 days.
- PF-02545920 (Cohort 3): Participants received PF-02545920 15 mg orally in a titrated manner over 18 days (titration scheme: 5 mg every 12 hours for 7 days, then 10 mg every 12 hours for 7 days, and then 15 mg every 12 hours for 4 days).
- Placebo (Cohort 3): Participants received placebo-matched to PF-02545920 tablets (Cohort 3) every 12 hours orally for 18 days.
Period: Overall Study
Arm/Group | PF-02545920 (Cohort 1) | PF-02545920 (Cohort 2) | Placebo (Cohorts 1 and 2) | PF-02545920 (Cohort 3) | Placebo (Cohort 3)
Started | 6 | 8 | 7 | 14 | 2
Completed | 6 | 8 | 7 | 12 | 2
Not Completed | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Groups:
- PF-02545920 (Cohort 1): Participants received PF-02545920 15 mg orally in a titrated manner over 10 days (titration scheme: 2 mg every 12 hours for 2 days, then 5 mg every 12 hours for 2 days, then 8 mg every 12 hours for 3 days, and then 15 mg every 12 hours for 3 days).
- Total: Total of all reporting groups
Arm/Group | PF-02545920 (Cohort 1) | PF-02545920 (Cohort 2) | Placebo (Cohorts 1 and 2) | PF-02545920 (Cohort 3) | Placebo (Cohort 3) | Total
Number analyzed (Participants) | 6 | 8 | 7 | 14 | 2 | 37
Age, Customized [Number; unit: participants]
  less than (<) 18 years | 0 | 0 | 0 | 0 | 0 | 0
  18-44 years | 1 | 7 | 1 | 5 | 2 | 16
  45-64 | 5 | 1 | 6 | 9 | 0 | 21
  Greater or equal to (>=) 65 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 0 | 0 | 3
  Male | 4 | 8 | 6 | 14 | 2 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Abbreviated Extrapyramidal Symptom Rating Scale (ESRS-A) Scores (Cohorts 1 and 2) at Day 10
Description: ESRS-A is a clinician rated scale consisting of 24 items to assess severity of extrapyramidal symptoms for following parameters: parkinsonism (10 items), dystonia (6 items), dyskinesia (6 items) and akathisia (2 items). Each item was scored on a 6-point scale (0=absent, 1=minimal, 2=mild, 3=moderate, 4=severe, 5=extreme). Additionally, 4 Clinical Global Impression of Severity (CGI-S) items were assessed on a 7-point scale (1=normal, not ill at all; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=extremely ill): CGI-S parkinsonism; CGI-S dystonia; CGI-S dyskinesia; CGI-S akathisia.
Time Frame: Day 0 (Baseline) up to Day 10
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-02545920 (Cohort 1) | PF-02545920 (Cohort 2) | Placebo (Cohorts 1 and 2)
Number analyzed (Participants) | 6 | 8 | 7
Units on a scale
  ESRS-A Parkinsonism | -0.2 (1.60) | -0.3 (0.46) | 0.1 (1.21)
  ESRS-A Dystonia | 0.0 (0.00) | 0.0 (0.00) | -0.1 (0.38)
  ESRS-A Dyskinesia | 0.0 (0.00) | 0.0 (0.00) | -0.1 (0.38)
  ESRS-A Akathisia | 0.0 (0.00) | 0.5 (0.93) | 0.0 (0.00)
  CGI-S Parkinsonism | 0.0 (0.63) | 0.0 (0.00) | 0.0 (0.58)
  CGI-S Dystonia | 0.0 (0.00) | 0.0 (0.00) | -0.1 (0.38)
  CGI-S Dyskinesia | 0.0 (0.00) | 0.0 (0.00) | -0.1 (0.38)
  CGI-S Akathisia | 0.0 (0.00) | 0.1 (0.35) | 0.0 (0.00)

2. Primary Outcome: Change From Baseline in ESRS-A Scores (Cohort 3) at Day 18
Description: ESRS-A is a clinician rated scale consisting of 24 items to assess severity of extrapyramidal symptoms for following parameters: parkinsonism (10 items), dystonia (6 items), dyskinesia (6 items) and akathisia (2 items). Each item is scored on a 6-point Likert scale (0=absent, 1=minimal, 2=mild, 3=moderate, 4=severe, 5=extreme). Additionally, 4 CGI-S items were assessed on a 7-point scale (1=normal, not ill at all; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=extremely ill): CGI-S parkinsonism; CGI-S dystonia; CGI-S dyskinesia; CGI-S akathisia.
Time Frame: Day 0 (Baseline) up to Day 18
Population: Safety analysis set included all participants who received at least 1 dose of study medication. Participants analyzed indicated number of evaluable participants.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-02545920 (Cohort 3) | Placebo (Cohort 3)
Number analyzed (Participants) | 12 | 2
Units on a scale
  ESRS-A Parkinsonism | 0.3 (1.50) | 0.0 (0.00)
  ESRS-A Dystonia | 0.0 (0.00) | 0.0 (0.00)
  ESRS-A Dyskinesia | 0.0 (0.00) | 0.0 (0.00)
  ESRS-A Akathisia | 0.6 (1.38) | 0.0 (0.00)
  CGI-S Parkinsonism | 0.2 (0.58) | 0.0 (0.00)
  CGI-S Dystonia | 0.0 (0.00) | 0.0 (0.00)
  CGI-S Dyskinesia | 0.0 (0.00) | 0.0 (0.00)
  CGI-S Akathisia | 0.3 (0.78) | 0.0 (0.00)

3. Primary Outcome: Number of Participants With Response to Columbia-Suicide Severity Rating Scale (C-SSRS) (Cohorts 1 and 2) at Baseline (Day 0)
Description: Data relevant to the assessment of suicidality was mapped to the Columbia-Classification Algorithm of Suicide Assessment (C-CASA) event codes. C-SSRS assessed whether participant experienced following: completed suicide (Event code 1), suicide attempt (Event code 2) (Response of "Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior (Event code 3) ("Yes" on "aborted attempt", "interrupted attempt", "preparatory acts or behavior"), suicidal ideation (Event code 4) ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act/some intent to act without specific plan or with specific plan and intent), self-injurious behavior, no suicidal intent (Event code 7) ("Yes" on "Has participant engaged in non-suicidal self-injurious behavior"). Number of participants with "Yes" response for above mentioned categories were assessed.
Time Frame: Day 0 (Baseline)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-02545920 (Cohort 1) | PF-02545920 (Cohort 2) | Placebo (Cohorts 1 and 2)
Number analyzed (Participants) | 6 | 8 | 7
Participants
  C-CASA Event Code 1 | 0 | 0 | 0
  C-CASA Event Code 2 | 0 | 0 | 0
  C-CASA Event Code 3 | 0 | 0 | 0
  C-CASA Event Code 4 | 0 | 0 | 0
  C-CASA Event Code 7 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Response to C-SSRS (Cohorts 1 and 2) at Day 11
Description: Data relevant to the assessment of suicidality was mapped to the C-CASA event codes. C-SSRS assessed whether participant experienced following: completed suicide (Event code 1), Suicide attempt (Event code 2) (Response of "Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior (Event code 3) ("Yes" on "aborted attempt", "interrupted attempt", "preparatory acts or behavior"), suicidal ideation (Event code 4) ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act/some intent to act without specific plan or with specific plan and intent), self-injurious behavior, no suicidal intent (Event code 7) ("Yes" on "Has participant engaged in non-suicidal self-injurious behavior"). Number of participants with "Yes" response for above mentioned categories were assessed.
Time Frame: Day 11
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | PF-02545920 (Cohort 1) | PF-02545920 (Cohort 2) | Placebo (Cohorts 1 and 2)
Number analyzed (Participants) | 5 | 8 | 6
Participants
  C-CASA Event Code 1 | 0 | 0 | 0
  C-CASA Event Code 2 | 0 | 0 | 0
  C-CASA Event Code 3 | 0 | 0 | 0
  C-CASA Event Code 4 | 0 | 0 | 0
  C-CASA Event Code 7 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Response to C-SSRS (Cohorts 1 and 2) at Follow-up (Any Day Between Day 17 and 20)
Description: as for outcome 4
Time Frame: Follow-up (any day between Day 17 and 20)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-02545920 (Cohort 1) | PF-02545920 (Cohort 2) | Placebo (Cohorts 1 and 2)
Number analyzed (Participants) | 6 | 8 | 7
Participants
  C-CASA Event Code 1 | 0 | 0 | 0
  C-CASA Event Code 2 | 0 | 0 | 0
  C-CASA Event Code 3 | 0 | 0 | 0
  C-CASA Event Code 4 | 0 | 0 | 0
  C-CASA Event Code 7 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Response to C-SSRS (Cohort 3) at Baseline (Day 0)
Description: as for outcome 4
Time Frame: Day 0 (Baseline)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-02545920 (Cohort 3) | Placebo (Cohort 3)
Number analyzed (Participants) | 14 | 2
Participants
  C-CASA Event Code 1 | 0 | 0
  C-CASA Event Code 2 | 0 | 0
  C-CASA Event Code 3 | 0 | 0
  C-CASA Event Code 4 | 0 | 0
  C-CASA Event Code 7 | 0 | 0

7. Primary Outcome: Number of Participants With Response to C-SSRS (Cohort 3) at Day 19
Description: as for outcome 4
Time Frame: Day 19
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | PF-02545920 (Cohort 3) | Placebo (Cohort 3)
Number analyzed (Participants) | 12 | 2
Participants
  C-CASA Event Code 1 | 0 | 0
  C-CASA Event Code 2 | 0 | 0
  C-CASA Event Code 3 | 0 | 0
  C-CASA Event Code 4 | 0 | 0
  C-CASA Event Code 7 | 0 | 0

8. Primary Outcome: Number of Participants With Response to C-SSRS (Cohort 3) at Follow-up (Any Day Between Day 26 and 29)
Description: as for outcome 4
Time Frame: Follow-up (any day between Day 26 and 29)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | PF-02545920 (Cohort 3) | Placebo (Cohort 3)
Number analyzed (Participants) | 12 | 2
Participants
  C-CASA Event Code 1 | 0 | 0
  C-CASA Event Code 2 | 0 | 0
  C-CASA Event Code 3 | 0 | 0
  C-CASA Event Code 4 | 0 | 0
  C-CASA Event Code 7 | 0 | 0

9. Primary Outcome: Number of Participants With Changes Since Screening in Physical Examination (Cohorts 1 and 2)
Description: A complete physical examination included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems was performed at Screening. The limited or abbreviated physical examination was focused on general appearance, the respiratory and cardiovascular systems, as well as towards assessment of subject reported symptoms and performed at other time points than Screening.
Time Frame: Screening up to Follow-up (any day between Day 17 and 20)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-02545920 (Cohort 1) | PF-02545920 (Cohort 2) | Placebo (Cohorts 1 and 2)
Number analyzed (Participants) | 6 | 8 | 7
Participants | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Changes Since Screening in Physical Examination (Cohort 3)
Description: as for outcome 9
Time Frame: Screening up to Follow-up (any day between Day 26 and 29)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-02545920 (Cohort 3) | Placebo (Cohort 3)
Number analyzed (Participants) | 14 | 2
Participants | 1 | 0

11. Primary Outcome: Number of Participants With Abnormal Neurological Examination Findings (Cohorts 1 and 2)
Description: The neurological examination included observation for cerebellar (intention) tremor and for non-cerebellar tremors (eg, resting or positional), finger-nose, heel-shin, Romberg, tandem walking, positional and gaze-evoked nystagmus.
Time Frame: Day 0 up to Follow-up (any day between Day 17 and 20)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-02545920 (Cohort 1) | PF-02545920 (Cohort 2) | Placebo (Cohorts 1 and 2)
Number analyzed (Participants) | 6 | 8 | 7
Participants | 2 | 0 | 1

12. Primary Outcome: Number of Participants With Abnormal Neurological Examination Findings (Cohort 3)
Description: as for outcome 11
Time Frame: Day 0 up to Follow-up (any day between Day 26 and 29)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-02545920 (Cohort 3) | Placebo (Cohort 3)
Number analyzed (Participants) | 14 | 2
Participants | 0 | 0

13. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) (Cohorts 1 and 2)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent were events between first dose of study drug and up to last subject visit that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: The time receiving the first dose of PF-02545920 or placebo through the last Follow-up (any day between Day 17 and 20)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-02545920 (Cohort 1) | PF-02545920 (Cohort 2) | Placebo (Cohorts 1 and 2)
Number analyzed (Participants) | 6 | 8 | 7
Participants | 5 | 5 | 3

14. Primary Outcome: Number of Participants With TEAEs (Cohort 3)
Description: as for outcome 13
Time Frame: The time receiving the first dose of PF-02545920/placebo through the last Follow-up (any day between Day 26 and 29)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-02545920 (Cohort 3) | Placebo (Cohort 3)
Number analyzed (Participants) | 14 | 2
Participants | 9 | 1

15. Primary Outcome: Number of Participants With Abnormal Clinical Laboratory Measurements (Cohorts 1 and 2)
Description: The total number of participants with laboratory test abnormalities without regard to baseline abnormality was assessed.
Time Frame: Day 0 (Baseline) up to Follow-up (any day between Day 17 and 20)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-02545920 (Cohort 1) | PF-02545920 (Cohort 2) | Placebo (Cohorts 1 and 2)
Number analyzed (Participants) | 6 | 8 | 7
Participants | 4 | 4 | 5

16. Primary Outcome: Number of Participants With Abnormal Clinical Laboratory Measurements (Cohort 3)
Description: The total number of participants with laboratory test abnormalities without regard to baseline abnormality was assessed.
Time Frame: Day 0 (Baseline) up to Follow-up (any day between Day 26 and 29)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | PF-02545920 (Cohort 3) | Placebo (Cohort 3)
Number analyzed (Participants) | 12 | 2
Participants | 11 | 0

17. Primary Outcome: Number of Participants With Vital Signs Data Meeting Criteria of Potential Clinical Concern (Cohorts 1 and 2)
Description: Vital signs included blood pressure (BP; supine and standing) and pulse rate. Vital signs criteria of potential clinical concern were 1), BP: systolic >=30 millimeters of mercury (mm Hg) change from baseline in same posture, systolic <90 mm Hg; diastolic >=20 mm Hg change from baseline in same posture, diastolic <50 mm Hg; 2), pulse rate (supine/sitting): <40 or greater than (>) 120 beats per minute (bpm); Standing: <40 or >140 bpm.
Time Frame: Day 0 (Baseline) up to Follow-up (any day between Day 17 and 20)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-02545920 (Cohort 1) | PF-02545920 (Cohort 2) | Placebo (Cohorts 1 and 2)
Number analyzed (Participants) | 6 | 8 | 7
Participants
  Supine systolic BP < 90 mm Hg | 1 | 1 | 0
  Standing systolic BP < 90 mm Hg | 0 | 1 | 0
  Increase in supine systolic BP >= 30 mm Hg | 1 | 1 | 1
  Increase in standing systolic BP >= 30 mm Hg | 1 | 0 | 0
  Increase in supine diastolic BP >= 20 mm Hg | 2 | 0 | 1
  Increase in standing diastolic BP >= 20 mm Hg | 1 | 0 | 1
  Decrease in supine systolic BP >= 30 mm Hg | 0 | 1 | 1
  Decrease in standing systolic BP >= 30 mm Hg | 0 | 1 | 2
  Decrease in supine diastolic BP >= 20 mm Hg | 0 | 3 | 1
  Decrease in standing diastolic BP >= 20 mm Hg | 1 | 2 | 1

18. Primary Outcome: Number of Participants With Vital Signs Data Meeting Criteria of Potential Clinical Concern (Cohort 3)
Description: Vital signs included BP (supine and standing) and pulse rate. Vital signs criteria of potential clinical concern were 1), BP: systolic >=30 mm Hg change from baseline in same posture, systolic <90 mm Hg; diastolic >=20 mm Hg change from baseline in same posture, diastolic <50 mm Hg; 2), pulse rate (supine/sitting): <40 or >120 bpm; Standing: <40 or >140 bpm.
Time Frame: Day 0 (Baseline) up to Follow-up (any day between Day 26 and 29)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | PF-02545920 (Cohort 3) | Placebo (Cohort 3)
Number analyzed (Participants) | 14 | 2
Participants
  Increase in supine systolic BP >= 30 mm Hg | 2 | 0
  Increase in standing systolic BP >= 30 mm Hg | 1 | 1
  Increase in supine diastolic BP >= 20 mm Hg | 1 | 0
  Decrease in supine systolic BP >= 30 mm Hg | 2 | 0
  Decrease in standing systolic BP >= 30 mm Hg | 6 | 1
  Decrease in supine diastolic BP >= 20 mm Hg | 3 | 0
  Decrease in standing diastolic BP >= 20 mm Hg | 7 | 1

19. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Criteria of Potential Clinical Concern (Cohorts 1 and 2)
Description: 12-lead ECG (triplicate) was performed on Day 0 and 12-lead ECG (singlet) was performed at other time points as specified in timeframe. ECG criteria of potential clinical concern were 1), PR interval: >=300 milliseconds (msec); >=25% increase when baseline was greater than (>) 200 msec; or increase >=50% when baseline was less than or equal to (<=) 200 msec; 2), QRS interval: >=140 msec; >=50% increase from baseline; 3), corrected QT interval (QTc interval): >=500 msec, QTc interval using Fridericia's formula (QTcF interval): absolute value >=450 - <480 msec(borderline), >=480 msec (prolonged); absolute change 30 - <60 (borderline), >=60 msec (prolonged).
Time Frame: Day 0 (Baseline) up to Day 10
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Groups:
- PF-02545920 (Cohort 1): Participants received PF-02545920 15 mg orally in a titrated manner over 18 days (titration scheme: 5 mg every 12 hours for 7 days, then 10 mg every 12 hours for 7 days, and then 15 mg every 12 hours for 4 days).
Arm/Group | PF-02545920 (Cohort 1) | PF-02545920 (Cohort 2) | Placebo (Cohorts 1 and 2)
Number analyzed (Participants) | 6 | 8 | 7
Participants | 0 | 0 | 0

20. Primary Outcome: Number of Participants With ECG Data Meeting Criteria of Potential Clinical Concern (Cohort 3)
Description: 12-lead ECG (triplicate)was performed on Day 0 and 12-lead ECG (singlet) was performed at other time points as specified in timeframe. ECG criteria of potential clinical concern were 1), PR interval: >=300 msec; >=25% increase when baseline >200 msec; or increase >=50% when baseline <=200 msec; 2), QRS interval: >=140 msec; >=50% increase from baseline; 3), QTc interval: >=500 msec, QTcF interval: absolute value >=450 - <480 msec (borderline), >=480 msec (prolonged); absolute change 30 - <60 (borderline), >=60 msec (prolonged).
Time Frame: Screening up to Day 18
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-02545920 (Cohort 3) | Placebo (Cohort 3)
Number analyzed (Participants) | 14 | 2
participants | 0 | 0

21. Primary Outcome: Sparse Pharmacokinetic (PK) Sampling for Population PK Analysis: PF-02545920 Concentration at 0 Hour (Predose) on Day 10 (Cohorts 1 and 2)
Time Frame: 0 hour (predose) on Day 10
Population: PK concentration population included all enrolled participants treated who had at least 1 measurable concentration.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | PF-02545920 (Cohort 1) | PF-02545920 (Cohort 2)
Number analyzed (Participants) | 6 | 8
nanogram/milliliter (ng/mL) | 45.07 (27.560) | 40.25 (31.465)

22. Primary Outcome: Sparse PK Sampling for Population PK Analysis: PF-02545920 Concentration at 25 Minutes (Post Dose) on Day 10 (Cohorts 1 and 2)
Time Frame: 25 minutes (post dose) on Day 10
Population: PK concentration population included all enrolled participants treated who had at least 1 measurable concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-02545920 (Cohort 1) | PF-02545920 (Cohort 2)
Number analyzed (Participants) | 6 | 8
ng/mL | 116.8 (72.996) | 138.3 (106.99)

23. Primary Outcome: Sparse PK Sampling for Population PK Analysis: PF-02545920 Concentration at 1 Hour 30 Minutes (Post Dose) on Day 10 (Cohorts 1 and 2)
Time Frame: 1 hour 30 minutes (post dose) on Day 10
Population: PK concentration population included all enrolled participants treated who had at least 1 measurable concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-02545920 (Cohort 1) | PF-02545920 (Cohort 2)
Number analyzed (Participants) | 6 | 8
ng/mL | 154.0 (48.248) | 151.1 (64.913)

24. Primary Outcome: Sparse PK Sampling for Population PK Analysis: PF-02545920 Concentration at 5 Hours (Post Dose) on Day 10 (Cohorts 1 and 2)
Time Frame: 5 hours (post dose) on Day 10
Population: PK concentration population included all enrolled participants treated who had at least 1 measurable concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-02545920 (Cohort 1) | PF-02545920 (Cohort 2)
Number analyzed (Participants) | 6 | 8
ng/mL | 62.38 (31.441) | 59.15 (33.294)

25. Primary Outcome: Sparse PK Sampling for Population PK Analysis: PF-02545920 Concentration at 24 Hours (Post Dose) on Day 10 (Cohorts 1 and 2)
Time Frame: 24 hours (post dose) on Day 10
Population: PK concentration population included all enrolled participants treated who had at least 1 measurable concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-02545920 (Cohort 1) | PF-02545920 (Cohort 2)
Number analyzed (Participants) | 5 | 8
ng/mL | 24.16 (21.032) | 21.11 (21.859)

26. Primary Outcome: Sparse PK Sampling for Population PK Analysis: PF-02545920 Concentration at 0 Hour (Predose) on Day 18 (Cohort 3)
Time Frame: 0 hour (predose) on Day 18
Population: PK concentration population included all enrolled participants treated who had at least 1 measurable concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-02545920 (Cohort 3)
Number analyzed (Participants) | 12
ng/mL | 42.71 (24.256)

27. Primary Outcome: Sparse PK Sampling for Population PK Analysis: PF-02545920 Concentration at 25 Minutes (Post Dose) on Day 18 (Cohort 3)
Time Frame: 25 minutes (post dose) Day 18
Population: PK concentration population included all enrolled participants treated who had at least 1 measurable concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-02545920 (Cohort 3)
Number analyzed (Participants) | 12
ng/mL | 156.1 (92.032)

28. Primary Outcome: Sparse PK Sampling for Population PK Analysis: PF-02545920 Concentration at 1 Hour 30 Minutes (Post Dose) on Day 18 (Cohort 3)
Time Frame: 1 hour 30 minutes (post dose) on Day 18
Population: PK concentration population included all enrolled participants treated who had at least 1 measurable concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-02545920 (Cohort 3)
Number analyzed (Participants) | 12
ng/mL | 156.4 (53.842)

29. Primary Outcome: Sparse PK Sampling for Population PK Analysis: PF-02545920 Concentration at 5 Hours (Post Dose) on Day 18 (Cohort 3)
Time Frame: 5 hours (post dose) on Day 18
Population: PK concentration population included all enrolled participants treated who had at least 1 measurable concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-02545920 (Cohort 3)
Number analyzed (Participants) | 12
ng/mL | 61.30 (23.764)

30. Primary Outcome: Sparse PK Sampling for Population PK Analysis: PF-02545920 Concentration at 24 Hours (Post Dose) on Day 18 (Cohort 3)
Time Frame: 24 hours (post dose) on Day 18
Population: PK concentration population included all enrolled participants treated who had at least 1 measurable concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-02545920 (Cohort 3)
Number analyzed (Participants) | 12
ng/mL | 20.85 (13.798)

ADVERSE EVENTS:
Time Frame: From the time the subject had taken at least 1 dose of study treatment through last subject visit. For serious AEs (SAEs), the time began from the subject provided informed consent through 28 calendar days post last administration of study drug.
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-02545920 (Cohort 1) | PF-02545920 (Cohort 2) | Placebo (Cohorts 1 and 2) | PF-02545920 (Cohort 3) | Placebo (Cohort 3)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/7 | 0/14 | 0/2
Other Adverse Events (participants affected / at risk) | 5/6 | 5/8 | 3/7 | 9/14 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-02545920 (Cohort 1) (N=6) | PF-02545920 (Cohort 2) (N=8) | Placebo (Cohorts 1 and 2) (N=7) | PF-02545920 (Cohort 3) (N=14) | Placebo (Cohort 3) (N=2)
Blepharospasm (Eye disorders) | 0 | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Orthostatic heart rate response increased (Investigations) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Akathisia (Nervous system disorders) | 1 | 3 | 0 | 3 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dystonia (Nervous system disorders) | 1 | 2 | 0 | 1 | 0
Extrapyramidal disorder (Nervous system disorders) | 1 | 0 | 0 | 3 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 4 | 0
Oromandibular dystonia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 5 | 3 | 0 | 7 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.